CLINICAL TRIAL: NCT06528678
Title: Visual Outcomes and Patient Satisfaction Results After Implantation of a Monofocal Intraocular Lens Designed for Monovision
Brief Title: Patients Outcomes of a Monofocal Intraocular Lens Designed for Monovision
Status: Completed | Type: Observational
Sponsor: Clinica Baviera (Other)
Responsible Party: Sponsor
Other Study IDs: LIO_EMV21
Record Dates: First submitted 2024-07-22; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cataract
Keywords: IOL; Monovision; Patient satisfaction
MeSH Terms: conditions — Cataract; Patient Satisfaction | interventions — Lenses, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- EMV monovision: Cataract surgery with EMV IOL
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Lens exchange with an intraocular lens

SUMMARY:
The rationale for this observational study of a CE-marked lens is to prospectively assess the performance, safety, and patient satisfaction in a group of subjects undergoing cataract surgery with bilateral implantation of the RayOne EMV in a monovision configuration. In order to increase the evidence collected from real-world clinical data we are running a multicentre clinical study in several clinics of the Baviera Ophthalmological Group.

Study design: prospective, observational, non-comparative.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Availability to complete follow-up examinations up to 6 months after surgery
* Cataract for which removal by phacoemulsification and subsequent IOL implantation was planned
* CDVA was expected to be better than 20/30 (+0.18 logMAR) after IOL implantation
* IOL power calculated in the range of +10.0 to +30.0 D
* Corneal astigmatism < 1.50 D
* Candidate for refractive surgery in monovision configuration

Exclusion Criteria:

* Women who were pregnant, nursing or planning to become pregnant during the study
* Difficulty for cooperation
* Inability to provide informed consent
* Concurrent participation in another investigational drug or device
* History of ocular trauma
* Previous intraocular or corneal surgery
* Presence of ocular pathologies
* Subjects with diagnosed degenerative visual disorders that were predicted to cause future acuity losses to a level of 20/30 or worse
* Subjects who may be expected to require retinal laser treatment
* Other eye condition that in the opinion of the investigator prevents the subject's participation in the study.
* Any other condition that may be contraindicated according to the IOL Instructions for Use.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cataract surgery at Clinica Baviera and implanted bilaterally with advanced monofocal intraocular lenses (RayOne EMV) with monovision configuration. The study population will comprise men and women aged 21 years or older and with an preoperative corneal astigmatism < 1.50 D.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Visual acuity | One month postoperative
  Visual acuity was measured using standard clinical charts
Defocus curve | One month postoperative
  Defocus curve was measured using standard clinical charts
Patient Satisfaction | One month postoperative
  Patient satisfaction was measured using the Cataract Assessment Patient Questionnaire 9 Short Form (Catquest 9SF) from 1 to 5, being 1 major difficulties and 5 cannot decide

SECONDARY OUTCOMES:
Safety of the device | Surgery, first follow-up visit (1-month) and second follow-up visit (6-months)
  Safety of the device was measured in terms of the frequency of adverse events related to the device
Quality of vision | One month postoperative
  Quality of vision was measured using a self-administered questionnaire developed at Clinica Baviera to assess patient satisfaction regarding night vision, from 1 to 4 being 1 the maximun score and 4 the worst score

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Baviera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Llovet-Rausell A, Navalon-Tortosa J, Druchkiv V, Coloma-Bockos J, Moya-Roca J, Llovet-Osuna F. Patient satisfaction and quality of vision after bilateral implantation of enhanced monofocal IOL and mini-monovision: a prospective study. Eye Vis (Lond). 2025 Jun 16;12(1):23. doi: 10.1186/s40662-025-00439-z. PMID 40524216